CLINICAL TRIAL: NCT03935724
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Delayed Start Phase II/III Study to Assess the Efficacy and Safety of Neuro-Cells in (Sub)Acute Spinal Cord Injury Patients
Brief Title: Stem Cells in Spinal Cord Injury
Acronym: SCI2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuroplast (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A2017SCI03
Record Dates: First submitted 2019-04-23; First posted 2019-05-02 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Spinal Cord Injuries; Acute Spinal Cord Injury; Paraplegia, Spinal; Paraplegia; Traumatic
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Intervention Model Description: Patients are randomized into two groups. First groups receives Neuro-cells, second group receives placebo. After six months second group also receives Neuro-cells. This happens in phase 2 and is repeated in phase 3. Therefore there are 4 groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties are masked (except for the care provider administering placebo of Neuro-cells). Unmasking will occur after six months when the placebo group receives Neuro-cells.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1A Intervention group 8 patients (Experimental): Neuro-Cells treatment at day 1-2 (= 6-10 weeks after TSCI incident). N=8
  Interventions: Biological: Neuro-Cells
- 1B Placebo group 8 patients (Placebo Comparator): Placebo treatment at day 1-2 (= 6-10 weeks after TSCI incident) Neuro-Cells treatment at day 181-182 (= 32-34 weeks after TSCI incident) N=8
  Interventions: Biological: Neuro-Cells
- 2A Intervention group 27 patients (Experimental): Neuro-Cells treatment at day 1-2 (= 6-10 weeks after TSCI incident) N=27
  Interventions: Biological: Neuro-Cells
- 2B Placebo group 27 patients (Placebo Comparator): Placebo treatment at day 1-2 (= 6-10 weeks after TSCI incident) Neuro-Cells treatment at day 181-182 (= 32-34 weeks after TSCI incident) N=27
  Interventions: Biological: Neuro-Cells

INTERVENTIONS:
Biological: Neuro-Cells — Neuro-Cells is an autologous fresh stem cells containing product which modulates the secondary inflammation following a TSCI, reduces apoptosis (cell death) in the injured spinal cord, reduces scar tissue formation in the damaged spinal cord and creates a cell regenerative environment in the injured spinal cord.

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled and delayed-start phase II/III clinical study.

DETAILED DESCRIPTION:
Phase II of the study focuses on establishing the safety and efficacy of the fist-in-human administration of Neuro-Cells. In phase III efficacy and safety will be further investigated. Enrollment in phase III of the study will automatically start once all patients have been enrolled and treated in phase II. The recruitment period is estimated at respectively 6 months for both the Phase II and Phase III.

Phase II starts with the enrollment of 16 evaluable patients, randomly divided in two groups of 8 evaluable patients each. After an interim intervention analysis, the phase II study expands into a phase III study, requiring the recruitment of 54 additional evaluable patients. Patients recruited for the phase III part will be randomly divided in two groups of 27 evaluable patients each. Details on the planned analyses can be found in section 8 'Statistical Analysis'.

Both the phase II and phase III part of the trial have a similar setup which includes a screening period (1 - 2 days), a randomization, a treatment period of 1 or 2 days and a total follow-up period of 1 year.

All patients undergo a BM harvesting at the start of their participation in the study and will undergo three LPs, performed to administer Neuro-Cells or placebo and/or to collect CSF for research purposes. Neuro-Cells and placebo are both administered as a single dose by an 'unblinded physician'. This physician is different from the 'blinded Investigators and study nurses' responsible for patient selection and follow-up. This study set-up allows to maintain a double-blind status of the patients and the Investigators responsible for the patients' evaluation throughout the first six months of both studies. This is because, approximately six months after the time of inclusion, the patients assigned to the placebo group will undergo a second BM harvesting and will also receive Neuro-Cells. All patients are followed up until approximately one year after the time of inclusion. All patients will have been treated with Neuro-Cells and will have completed follow-up for at least 6 months post-treatment. Patient recruitment, randomization and blinding, and the primary and secondary objectives are identical in the phase II and the phase III part of the study. The study is completed when the last patient finishes his/her last visit, approximately one year after the time of inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 - 65 years
* Complete (AIS grade A) or incomplete (AIS grade B or C) TSCI (ISNCSCI-assessed) at time of randomization
* Randomization can be done within 6-10 weeks after the TSCI incident
* Level of injury between C4 to T12
* Voluntary signed informed consent by patients and Investigator before any trial-related procedures are performed

Exclusion Criteria:

* SCI AIS grade D or E at the start of enrolment
* Level of SCI above C4 or below T12
* Positive HIV, hepatitis B or C serology
* Positive Lues test
* Total Nuclear Cell (TNC) count < 1x109 TNC
* Cancer, brain injury, disturbed consciousness, signs/symptoms of neurodegenerative disorder (e.g. stroke, amyotrophic lateral sclerosis, multiple sclerosis etc), diabetes mellitus type 1, renal or cardiac insufficiency based on anamnesis history and at the investigator's discretion
* Patients suffering from respiratory issues that cannot breathe on their own 24/7
* Any concomitant treatment or medication that interferes with the conduct of the trial, such as immune-suppressive medication or other medication (especially methotrexate, cyclosporine, and corticosteroids have to be avoided) known to interact with the anti- inflammatory and immune-modulative actions of stem cells (non-steroid anti- inflammatory drugs (NSAIDs) are allowed)
* Abuse of alcohol (daily consumption of more than 2 units of alcohol containing drinks) or illicit drugs (e.g. heroin, cocaine, XTC)
* Individuals that belong to vulnerable population groups
* Females with childbearing potential without using adequate birth control methods, and/or being pregnant or in the lactation period
* Participation in any clinical trial (with exemption of descriptive studies with questionnaires and no active intervention) within the previous 30 days before enrolment, or simultaneous participation in such trial
* Patients with extreme comorbidity before or after the TSCI are excluded at discretion of the PI
* Patients who are unable to comply with the requirements of this clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Physical changes after intrathecal intervention with Neuro-Cells | 9 months
  At approx. 3 months after intrathecal intervention with Neuro-Cells (day 90 for the patients treated 6-10 weeks after the TSCI incident and day 270 for the patients treated at 32-34 weeks after the TSCI incident) a physical examination (checklist) will be done
Increase of motor scores after intrathecal invervention with Neuro-Cells | 6 months
  Increase in the ISNCSCI motor scores with additional 5 points from baseline (visit 2) at 6 months after the intrathecal intervention (day 180) in patients treated with Neuro-Cells

SECONDARY OUTCOMES:
Increase of motor scores after late administration of Neuro-Cells | 12 months
  Increase in the ISNCSCI motor scores with additional 5 points from baseline (visit 5) at 6 months after the intrathecal intervention (day 360) in patients treated with Neuro-Cells 32 to 34 weeks after the TSCI incident as compared to placebo treated patients
Change in autonomic and sensoric neurological dysfunctionafter intrathecal invervention with Neuro-Cells | 12 months
  The American Spinal Injury Association (ASIA) Impairment Scale involves both a Motor and Sensory examination for each side of the body (left/right).
  The Sensory examination involves 'light touch' and 'pinprick' for each dermatome (28) on both sides of the body (total 56). A score of 0, 1 or 2 can be given to each dermatome resulting in a total max. of 112 points.
  The Motor level is determined by examining the muscle function within each of the 10 myotomes on each side of the body (20 myotomes in total). A score ranging from 1 to 5 can be given resulting in a maximum score of 100.
  The higher the value, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Oliviero, MD, Principal Investigator — Hospital Nacional de Parapléjicos de Toledo; Fin Biering-Soerensen, MD, Principal Investigator — Righospitalet
Locations (2):
- Rigshospitalet, Copenhagen, Denmark
- Hospital Nacional de Parapléjicos, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website Neuroplast — https://www.neuroplast.com/